CLINICAL TRIAL: NCT02456831
Title: Efficacy of Soy Formula Feedings in Healthy, Term Infants
Brief Title: Soy Formula Feedings in Healthy, Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AE58
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control Infant Formula (Active Comparator): Ready-to-Feed (RTF) Soy Infant Formula
  Interventions: Other: Active Comparator: Control Infant Formula
- Experimental Infant Formula 1 (Experimental): Experimental Ready-to-Feed Soy Formula
  Interventions: Other: Experimental Infant Formula 1
- Experimental Infant Formula 2 (Experimental): Experimental Ready-to-Feed Soy Formula
  Interventions: Other: Experimental Infant Formula 2
- Experimental Infant Formula 3 (Experimental): Experimental Ready-to-Feed Soy Formula
  Interventions: Other: Experimental Infant Formula 3

INTERVENTIONS:
Other: Experimental Infant Formula 1 — method A phytate reduction and 5% protein hydrolysis
  Arms: Experimental Infant Formula 1
Other: Experimental Infant Formula 2 — method A phytate reduction and 10% protein hydrolysis
  Arms: Experimental Infant Formula 2
Other: Experimental Infant Formula 3 — method B phytate reduction and 5% protein hydrolysis
  Arms: Experimental Infant Formula 3
Other: Active Comparator: Control Infant Formula — Ready-to-Feed (RTF) Soy Infant Formula
  Arms: Control Infant Formula

SUMMARY:
This study evaluates the GI tolerance and acceptability of soy formulas fed to healthy term infants with reported intolerance to a milk-based formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants believed by their parents and/or physicians to be experiencing symptoms of cow's milk formula intolerance and who had not previously consumed a soy-based formula (Intervention subjects).
* Health infants reported to be tolerating a milk-based formula (Cohorts).
* Infants considered full-term, 2 to 9 weeks of age with a birth-weight above the 5th percentile (NCHS).

Ages: 2 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 1992-12; Primary Completion 1994-06 (Actual); Study Completion 1994-06 (Actual)

PRIMARY OUTCOMES:
Stool Characteristics Questionnaire | Change from Baseline (Study Day 1) to Study Day 15
  stool number, consistency, and color

SECONDARY OUTCOMES:
Formula Intake | Change from Baseline (Study Day 1) to Study Day 15
  volume consumed
Gastrointestinal Tolerance Questionnaire | Change from Baseline (Study Day 1) to Study Day 15
  Incidence of spit up and vomiting
Weight | Change from Baseline (Study Day 1) to Study Day 15
  weight and weight gain

CONTACTS AND LOCATIONS:
Overall Officials: John Lasekan, MBA, PhD, CCRP, Study Chair — Abbott Nutrition
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Dreyer Clinic, Aurora, Illinois
  - T&W Research, Owensboro, Kentucky
  - Park Nicollet Medical Foundation, Minneapolis, Minnesota
  - Clinical Studies, Inc, Canton, Ohio
  - Research Memphis, Memphis, Tennessee
  - Child Care Associates, San Antonio, Texas